CLINICAL TRIAL: NCT02597127
Title: A Placebo-controlled, Double-blind, Randomized Trial to Compare the Effect of Different Doses of ALN-PCSSC Given as Single or Multiple Subcutaneous Injections in Subjects With High Cardiovascular Risk and Elevated LDL-C
Brief Title: Trial to Evaluate the Effect of ALN-PCSSC Treatment on Low Density Lipoprotein Cholesterol (LDL-C)
Acronym: ORION-1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MDCO-PCS-15-01
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Results first posted 2019-05-17 (Actual); Last update posted 2019-05-17 (Actual); Status verified 2019-04

CONDITIONS: Atherosclerotic Cardiovascular Disease; Familial Hypercholesterolemia; Diabetes
MeSH Terms: conditions — Atherosclerosis; Hyperlipoproteinemia Type II; Diabetes Mellitus | interventions — ALN-PCS; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- ALN-PCSSC 200 mg (bi-annual dosing) (Experimental): ALN-PCSSC 200 milligram (mg) SC administration once at Day 1
  Interventions: Drug: ALN-PCSSC
- ALN-PCSSC 300 mg (bi-annual dosing) (Experimental): ALN-PCSSC 300 mg SC administration once at Day 1
  Interventions: Drug: ALN-PCSSC
- ALN-PCSSC 500 mg (bi-annual dosing) (Experimental): ALN-PCSSC 500 mg SC administration once at Day 1
  Interventions: Drug: ALN-PCSSC
- Normal Saline (bi-annual dosing) (Placebo Comparator): Saline SC administration once at Day 1
  Interventions: Drug: Normal Saline
- ALN-PCSSC 100 mg (quarterly dosing) (Experimental): ALN-PCSSC 100 mg SC administration twice at Day 1 and Day 90
  Interventions: Drug: ALN-PCSSC
- ALN-PCSSC 200 mg (quarterly dosing) (Experimental): ALN-PCSSC 200 mg SC administration twice at Day 1 and Day 90
  Interventions: Drug: ALN-PCSSC
- ALN-PCSSC 300 mg (quarterly dosing) (Experimental): ALN-PCSSC 300 mg SC administration twice at Day 1 and Day 90
  Interventions: Drug: ALN-PCSSC
- Normal Saline (quarterly dosing) (Placebo Comparator): Saline SC administration twice at Day 1 and Day 90
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: ALN-PCSSC — ALN-PCSSC is a small interfering ribonucleic acid (RNA) that inhibits PCSK9 synthesis and is given as SC injections
  Other Names: PCSK9 synthesis inhibitor; Inclisiran
  Arms: ALN-PCSSC 100 mg (quarterly dosing); ALN-PCSSC 200 mg (bi-annual dosing); ALN-PCSSC 200 mg (quarterly dosing); ALN-PCSSC 300 mg (bi-annual dosing); ALN-PCSSC 300 mg (quarterly dosing); ALN-PCSSC 500 mg (bi-annual dosing)
Drug: Normal Saline — Saline (sterile, normal, 0.9%) solution given as SC injections
  Arms: Normal Saline (bi-annual dosing); Normal Saline (quarterly dosing)

SUMMARY:
This study is a Phase II, placebo-controlled, double-blind, randomized trial in 480 participants with atherosclerotic cardiovascular disease (ASCVD) or ASCVD-risk equivalents (for example, diabetes and familial hypercholesterolemia) and elevated LDL-C despite maximum tolerated dose of LDL-C lowering therapies to evaluate the efficacy, safety, and tolerability of ALN-PCSSC injection(s).

DETAILED DESCRIPTION:
Participants will be screened and 480 eligible participants will be randomized: 60 participants per each of six ALN-PCSSC dose groups plus 120 participants total across the placebo groups (20 participants each to match each of the six drug dose groups). Treatment allocation will be stratified by country and by current use of statins or other lipid-modifying therapies. Each participant will receive either one or two injections on Day 1 or a single injection on Day 1 and on Day 90 of blinded ALN-PCSSC or placebo.

Formation of anti-drug antibodies (ADA) will be assessed on Day 1 (prior to and 4 hours after the injection) and on Days 30, 60, 90, 120, 150, 180 (Days 150 and 180 only in participants who receive a second dose of study drug), and 210 or until any ADA response becomes negative within the study duration.

The independent Data Monitoring Committee (DMC) will review safety data beginning after the first 40 participants receive the first injection of ALN-PCSSC or placebo and complete the Day 14 follow-up visit. Thereafter, the DMC will review safety data every 2 months until the end of the trial. A recommendation may be taken to stop or amend the study at any of these reviews.

On Day 1, all eligible participants will be randomized and receive the first subcutaneous (SC) administration of ALN-PCSSC or placebo. After the first study drug administration, the participant will be observed in the clinic for at least 4 hours post injection before being discharged. Participants will return at Day 14 and then at monthly intervals for 6 months. Participants randomized to receive a second dose of study drug will receive the second injection of ALN-PCSSC or placebo at the Day 90 visit.

Efficacy assessments will include the measurement of the effects of ALN-PCSSC on levels of LDL-C lipids and lipoproteins including total cholesterol (TC), triglycerides, high-density lipoprotein cholesterol (HDL-C), non-HDL-C, very low-density lipoprotein (VLDL), apolipoprotein A1 (Apo-AI), apolipoprotein B (Apo-B), lipoprotein (a) [Lp(a)], C-reactive protein (CRP), and proprotein convertase subtilisin/kexin type 9 (PCSK9).

End of study (EOS) evaluations will be conducted at the EOS visit (Day 210). The expected duration of the participants' involvement in the study will be approximately 374 days, which includes screening, study drug administration, the course of single or multiple injections, and the follow-up period to Day 360.

Participants completing the study to Day 210 will be given the opportunity to enroll in a separate long-term extension study. Any participants in whom LDL-C levels have not returned to >80% of baseline values will continue to be followed as part of this study until either this level has been reached or until a maximum of Day 360, at which point they will be given the opportunity to enroll in the long-term extension study. At each visit, LDL-C levels, adverse events, serious adverse events, concomitant medications, and safety laboratory assessments will be collected.

Objectives:

Primary:

To evaluate the effect of ALN-PCSSC treatment on LDL-C levels at Day 180.

Secondary:

To evaluate the effect of ALN-PCSSC on the following:

* LDL-C at Day 90
* LDL-C levels at other time points
* PCSK9 levels over time
* Other lipids, lipoproteins, apolipoproteins
* Proportion of participants achieving pre-specified global lipid guidelines
* Individual responsiveness to different doses
* Duration of lipid-lowering effect of different doses
* Safety and tolerability profile of ALN-PCSSC

Exploratory:

To collect/evaluate the effect of ALN-PCSSC on the following:

* Cardiovascular (CV) events such as CV death, non-fatal myocardial infarction, resuscitated cardiac arrest and non-fatal stroke (ischemic and hemorrhagic)
* Evaluation of ADA for the investigational product

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants ≥18 years of age.
2. History of ASCVD or ASCVD-risk equivalents (symptomatic atherosclerosis, Type 2 diabetes, familial hypercholesterolemia, including participants whose 10-year risk of a CV event assessed by Framingham Risk Score (Framingham Risk Score >20%) or equivalent has a target LDL-C of <100 mg/deciliter [dL]).
3. Serum LDL-C ≥1.8 millimole (mmol)/liter (L) (≥70 mg/dL) for ASCVD participants or ≥2.6 mmol/L (≥100 mg/dL) for ASCVD-risk equivalent participants at screening.
4. Fasting triglyceride <4.52 mmol/L (<400 mg/dL) at screening.
5. Calculated glomerular filtration rate 30 mL/min or higher by estimated glomerular filtration rate (eGFR) using standardized local clinical methodology.
6. Participants on statins should be receiving a maximally tolerated dose (investigator's discretion).
7. Participants on lipid-lower therapies (such as statin and/or ezetimibe) should be on a stable dose for ≥30 days before screening with no planned medication or dose change during study participation.
8. Willing and able to give informed consent before initiation of any study-related procedures and willing to comply with all required study procedures.

Exclusion Criteria:

1. Any uncontrolled or serious disease, or any medical or surgical condition, that may either interfere with participation in the clinical study, and/or put the participant at significant risk (according to investigator's [or delegate] judgment) if he/she participates in the clinical study.
2. An underlying known disease, or surgical, physical, or medical condition that, in the opinion of the investigator (or delegate), might interfere with interpretation of the clinical study results.
3. New York Heart Association (NYHA) class II, III, or IV heart failure or last known left ventricular ejection fraction <30%.
4. Cardiac arrhythmia within 3 months prior to randomization that is not controlled by medication or via ablation.
5. Any history of hemorrhagic stroke.
6. Major adverse cardiac event within 6 months prior to randomization.
7. Uncontrolled severe hypertension: systolic blood pressure >180 millimeters of mercury (mmHg) or diastolic blood pressure >110 mmHg prior to randomization despite anti-hypertensive therapy.
8. Poorly controlled Type 2 diabetes, such as, glycated hemoglobin A1c (HbA1c)>10.0% prior to randomization.
9. Active liver disease defined as any known current infectious, neoplastic, or metabolic pathology of the liver or unexplained alanine aminotransferase (ALT) or aspartate aminotransferase (AST) elevation >2x the upper limit of normal (ULN), or total bilirubin elevation >1.5x ULN at screening confirmed by a repeat measurement at least 1 week apart.
10. Serious comorbid disease in which the life expectancy of the participant is shorter than the duration of the trial (for example, acute systemic infection, cancer, or other serious illnesses). This includes all cancers with the exception of treated basal-cell carcinoma occurring >5 years before screening.
11. Females who are pregnant or nursing, or who are of childbearing potential and unwilling to use at least two methods of contraception (oral contraceptives, barrier methods, approved contraceptive implant, long-term injectable contraception, intrauterine device or tubal litigation) for the entire duration of the study. Women who are >2 years postmenopausal defined as ≥1 year since last menstrual period and if less than 55 years old with a negative pregnancy test within 24 hours of randomization or surgically sterile are exempt from this exclusion.
12. Males who are unwilling to use an acceptable method of birth control during the entire study period (such as, condom with spermicide).
13. Known history of alcohol and/or drug abuse within the last 5 years.
14. Treatment with other investigational medicinal products or devices within 30 days or five half˗lives, whichever is longer.
15. Use of other investigational medicinal products or devices during the course of the study.
16. Any condition that according to the investigator could interfere with the conduct of the study, such as but not limited to the following:

    * Inappropriate for this study, including participants who are unable to communicate or to cooperate with the investigator.
    * Unable to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study (including participants whose cooperation is doubtful due to drug abuse or alcohol dependency).
    * Unlikely to comply with the protocol requirements, instructions, and study-related restrictions (for example, uncooperative attitude, inability to return for follow-up visits, and improbability of completing the study).
    * Have any medical or surgical condition, which in the opinion of the investigator would put the participants at increased risk from participating in the study.
    * Involved with, or a relative of, someone directly involved in the conduct of the study.
    * Any known cognitive impairment (for example, Alzheimer's disease)
17. Previous or current treatment (within 90 days of screening) with monoclonal antibodies directed at PCSK9.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 501 (Actual)
Dates: Start 2016-01; Primary Completion 2017-06-07 (Actual); Study Completion 2017-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kausik K Ray, MD, Principal Investigator — Department of Public Health and Primary Care, Imperial College London, Reynolds Building
Locations (54):
- United States (8):
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Midwest Institute For Clinical Research, Indianapolis, Indiana
  - Mount Sinai Icahn School of Medicine, New York, New York
  - Metabolic And Atherosclerosis Research Center, Cincinnati, Ohio
  - Sterling Research Group, Cincinnati, Ohio
  - Wellmont CVA Heart Institute, Greeneville, Tennessee
  - Amarillo Heart Clinical Research Institute, Inc., Amarillo, Texas
  - National Clinical Research, Inc., Richmond, Virginia
- Canada (12):
  - St. Paul's Hospital, Vancouver, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Eastern Regional Health Authority, Patient Research Centre, St. John's, Newfoundland and Labrador
  - Brampton Research Associates, Brampton, Ontario
  - Lawson Health Research Institute, London, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - ECOGENE-21 Clinical Trials Center, Chicoutimi, Quebec
  - Clinic Sante Cardio MC, Montreal, Quebec
  - Institut de Recherches Cliniques de Montreal, Montreal, Quebec
  - Université Laval Quebec, Québec, Quebec
  - Clinique des maladies lipidique Quebec, Québec, Quebec
  - Centre intégré universitaire de santé et de services sociaux de l'Estrie - Centre hospitalier universitaire de Sherbrooke (CIUSSS de l'Estrie - CHUS), Sherbrooke, Quebec
- Germany (6):
  - Medical University Berlin, Berlin
  - Medical Center Essen, Essen
  - University Hospital Frankfurt, Frankfurt
  - University Heart Center Hamburg, Hamburg
  - Medical University Hospital Heidelberg, Internal medicine III, Heidelberg
  - Technical University Munich, German Heart Center, Munich
- Netherlands (14):
  - Amsterdam Medical Center, Amsterdam
  - Deventer Ziekenhuis, Deventer
  - Andromed Eindhoven, Eindhoven
  - Admiraal de Ruyter Hospital, Cardiology, Goes
  - Bethesda Diabetes Research Center, Hoogeveen
  - Medisch Centrum Gorecht, Hoogezand
  - VOC Hoorn, Hoorn
  - Leids Universitair Medisch Centrum (LUMC), Leiden
  - Andromed Rotterdam, Rotterdam
  - Haga Hospital, The Hague
  - Diakonessenhuis, Vascular Policlinic, Utrecht
  - UMC Utrecht, Utrecht
  - VieCurie Venlo, Cardiology, Venlo
  - Albert Schweitzer Hospital, Cardiology, Zwijndrecht
- United Kingdom (14):
  - Queen Elizabeth Hospital, University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Edinburgh Royal Infirmary, Edinburgh
  - The Royal Devon and Exeter NHS Trust, Exeter
  - Fowey River Practice, Fowey
  - Buckinghamshire NHS Trust, High Wycombe
  - Oak Tree Surgery, Liskeard
  - Royal Free Hospital, London
  - Central Manchester University Hospital NHS Foundation Trust, Manchester
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Freeman Hospital, Newcastle upon Tyne
  - The Alverton Practice, Penzance
  - Knowle House Surgery, Plymouth
  - Brannel Surgery, St Austell
  - Rame Medical Ltd (Rame Research), Torpoint
  - Worcestershire Acute NHS Trust, Worcester

REFERENCES:
- [Background] Abifadel M, Varret M, Rabes JP, Allard D, Ouguerram K, Devillers M, Cruaud C, Benjannet S, Wickham L, Erlich D, Derre A, Villeger L, Farnier M, Beucler I, Bruckert E, Chambaz J, Chanu B, Lecerf JM, Luc G, Moulin P, Weissenbach J, Prat A, Krempf M, Junien C, Seidah NG, Boileau C. Mutations in PCSK9 cause autosomal dominant hypercholesterolemia. Nat Genet. 2003 Jun;34(2):154-6. doi: 10.1038/ng1161. PMID 12730697
- [Background] Ashwell G, Morell AG. The role of surface carbohydrates in the hepatic recognition and transport of circulating glycoproteins. Adv Enzymol Relat Areas Mol Biol. 1974;41(0):99-128. doi: 10.1002/9780470122860.ch3. No abstract available. PMID 4609051
- [Background] Banerjee Y, Shah K, Al-Rasadi K. Effect of a monoclonal antibody to PCSK9 on LDL cholesterol. N Engl J Med. 2012 Jun 21;366(25):2425-6; author reply 2426. doi: 10.1056/NEJMc1204929. No abstract available. PMID 22716984
- [Background] Milazzo L, Antinori S. Effect of a monoclonal antibody to PCSK9 on LDL cholesterol. N Engl J Med. 2012 Jun 21;366(25):2425; author reply 2426. doi: 10.1056/NEJMc1204929. No abstract available. PMID 22716983
- [Background] Cholesterol Treatment Trialists' (CTT) Collaboration; Baigent C, Blackwell L, Emberson J, Holland LE, Reith C, Bhala N, Peto R, Barnes EH, Keech A, Simes J, Collins R. Efficacy and safety of more intensive lowering of LDL cholesterol: a meta-analysis of data from 170,000 participants in 26 randomised trials. Lancet. 2010 Nov 13;376(9753):1670-81. doi: 10.1016/S0140-6736(10)61350-5. Epub 2010 Nov 8. PMID 21067804
- [Background] Coelho T, Adams D, Silva A, Lozeron P, Hawkins PN, Mant T, Perez J, Chiesa J, Warrington S, Tranter E, Munisamy M, Falzone R, Harrop J, Cehelsky J, Bettencourt BR, Geissler M, Butler JS, Sehgal A, Meyers RE, Chen Q, Borland T, Hutabarat RM, Clausen VA, Alvarez R, Fitzgerald K, Gamba-Vitalo C, Nochur SV, Vaishnaw AK, Sah DW, Gollob JA, Suhr OB. Safety and efficacy of RNAi therapy for transthyretin amyloidosis. N Engl J Med. 2013 Aug 29;369(9):819-29. doi: 10.1056/NEJMoa1208760. PMID 23984729
- [Background] Cohen JC, Boerwinkle E, Mosley TH Jr, Hobbs HH. Sequence variations in PCSK9, low LDL, and protection against coronary heart disease. N Engl J Med. 2006 Mar 23;354(12):1264-72. doi: 10.1056/NEJMoa054013. PMID 16554528
- [Background] Davidson MH, Maki KC, Pearson TA, Pasternak RC, Deedwania PC, McKenney JM, Fonarow GC, Maron DJ, Ansell BJ, Clark LT, Ballantyne CM. Results of the National Cholesterol Education (NCEP) Program Evaluation ProjecT Utilizing Novel E-Technology (NEPTUNE) II survey and implications for treatment under the recent NCEP Writing Group recommendations. Am J Cardiol. 2005 Aug 15;96(4):556-63. doi: 10.1016/j.amjcard.2005.04.019. PMID 16098311
- [Background] Dias CS, Shaywitz AJ, Wasserman SM, Smith BP, Gao B, Stolman DS, Crispino CP, Smirnakis KV, Emery MG, Colbert A, Gibbs JP, Retter MW, Cooke BP, Uy ST, Matson M, Stein EA. Effects of AMG 145 on low-density lipoprotein cholesterol levels: results from 2 randomized, double-blind, placebo-controlled, ascending-dose phase 1 studies in healthy volunteers and hypercholesterolemic subjects on statins. J Am Coll Cardiol. 2012 Nov 6;60(19):1888-98. doi: 10.1016/j.jacc.2012.08.986. Epub 2012 Oct 17. PMID 23083772
- [Background] Elbashir SM, Harborth J, Lendeckel W, Yalcin A, Weber K, Tuschl T. Duplexes of 21-nucleotide RNAs mediate RNA interference in cultured mammalian cells. Nature. 2001 May 24;411(6836):494-8. doi: 10.1038/35078107. PMID 11373684
- [Background] Foley KA, Simpson RJ Jr, Crouse JR 3rd, Weiss TW, Markson LE, Alexander CM. Effectiveness of statin titration on low-density lipoprotein cholesterol goal attainment in patients at high risk of atherogenic events. Am J Cardiol. 2003 Jul 1;92(1):79-81. doi: 10.1016/s0002-9149(03)00474-0. No abstract available. PMID 12842255
- [Background] Foody JM, Sajjan SG, Hu XH, Ramey DR, Neff DR, Tershakovec AM, Tomassini JE, Wentworth C, Tunceli K. Loss of early gains in low-density lipoprotein cholesterol goal attainment among high-risk patients. J Clin Lipidol. 2010 Mar-Apr;4(2):126-32. doi: 10.1016/j.jacl.2010.01.007. Epub 2010 Feb 6. PMID 21122640
- [Background] ALN TTRSC-001; EudraCT 2012 004203 12
- [Background] ALN-TTRSC-002; EudraCT 2013 002856 33
- [Background] Geisbert TW, Hensley LE, Kagan E, Yu EZ, Geisbert JB, Daddario-DiCaprio K, Fritz EA, Jahrling PB, McClintock K, Phelps JR, Lee AC, Judge A, Jeffs LB, MacLachlan I. Postexposure protection of guinea pigs against a lethal ebola virus challenge is conferred by RNA interference. J Infect Dis. 2006 Jun 15;193(12):1650-7. doi: 10.1086/504267. Epub 2006 May 10. PMID 16703508
- [Background] Grundy SM, Cleeman JI, Merz CN, Brewer HB Jr, Clark LT, Hunninghake DB, Pasternak RC, Smith SC Jr, Stone NJ; National Heart, Lung, and Blood Institute; American College of Cardiology Foundation; American Heart Association. Implications of recent clinical trials for the National Cholesterol Education Program Adult Treatment Panel III guidelines. Circulation. 2004 Jul 13;110(2):227-39. doi: 10.1161/01.CIR.0000133317.49796.0E. PMID 15249516
- [Background] Hooper AJ, Marais AD, Tanyanyiwa DM, Burnett JR. The C679X mutation in PCSK9 is present and lowers blood cholesterol in a Southern African population. Atherosclerosis. 2007 Aug;193(2):445-8. doi: 10.1016/j.atherosclerosis.2006.08.039. Epub 2006 Sep 20. PMID 16989838
- [Background] Hooper AJ, Burnett JR. Anti-PCSK9 therapies for the treatment of hypercholesterolemia. Expert Opin Biol Ther. 2013 Mar;13(3):429-35. doi: 10.1517/14712598.2012.748743. Epub 2012 Dec 17. PMID 23240807
- [Background] Horton JD, Cohen JC, Hobbs HH. PCSK9: a convertase that coordinates LDL catabolism. J Lipid Res. 2009 Apr;50 Suppl(Suppl):S172-7. doi: 10.1194/jlr.R800091-JLR200. Epub 2008 Nov 19. PMID 19020338
- [Background] Judge AD, Bola G, Lee AC, MacLachlan I. Design of noninflammatory synthetic siRNA mediating potent gene silencing in vivo. Mol Ther. 2006 Mar;13(3):494-505. doi: 10.1016/j.ymthe.2005.11.002. Epub 2005 Dec 15. PMID 16343994
- [Background] Cholesterol Treatment Trialists' (CTT) Collaborators; Kearney PM, Blackwell L, Collins R, Keech A, Simes J, Peto R, Armitage J, Baigent C. Efficacy of cholesterol-lowering therapy in 18,686 people with diabetes in 14 randomised trials of statins: a meta-analysis. Lancet. 2008 Jan 12;371(9607):117-25. doi: 10.1016/S0140-6736(08)60104-X. PMID 18191683
- [Background] Morrissey DV, Lockridge JA, Shaw L, Blanchard K, Jensen K, Breen W, Hartsough K, Machemer L, Radka S, Jadhav V, Vaish N, Zinnen S, Vargeese C, Bowman K, Shaffer CS, Jeffs LB, Judge A, MacLachlan I, Polisky B. Potent and persistent in vivo anti-HBV activity of chemically modified siRNAs. Nat Biotechnol. 2005 Aug;23(8):1002-7. doi: 10.1038/nbt1122. Epub 2005 Jul 24. PMID 16041363
- [Background] Mousavi SA, Berge KE, Leren TP. The unique role of proprotein convertase subtilisin/kexin 9 in cholesterol homeostasis. J Intern Med. 2009 Dec;266(6):507-19. doi: 10.1111/j.1365-2796.2009.02167.x. PMID 19930098
- [Background] Nag SS, Daniel GW, Bullano MF, Kamal-Bahl S, Sajjan SG, Hu H, Alexander C. LDL-C goal attainment among patients newly diagnosed with coronary heart disease or diabetes in a commercial HMO. J Manag Care Pharm. 2007 Oct;13(8):652-63. doi: 10.18553/jmcp.2007.13.8.652. PMID 17970603
- [Background] Raal F, Scott R, Somaratne R, Bridges I, Li G, Wasserman SM, Stein EA. Low-density lipoprotein cholesterol-lowering effects of AMG 145, a monoclonal antibody to proprotein convertase subtilisin/kexin type 9 serine protease in patients with heterozygous familial hypercholesterolemia: the Reduction of LDL-C with PCSK9 Inhibition in Heterozygous Familial Hypercholesterolemia Disorder (RUTHERFORD) randomized trial. Circulation. 2012 Nov 13;126(20):2408-17. doi: 10.1161/CIRCULATIONAHA.112.144055. Epub 2012 Nov 5. PMID 23129602
- [Background] European Association for Cardiovascular Prevention & Rehabilitation; Reiner Z, Catapano AL, De Backer G, Graham I, Taskinen MR, Wiklund O, Agewall S, Alegria E, Chapman MJ, Durrington P, Erdine S, Halcox J, Hobbs R, Kjekshus J, Filardi PP, Riccardi G, Storey RF, Wood D; ESC Committee for Practice Guidelines (CPG) 2008-2010 and 2010-2012 Committees. ESC/EAS Guidelines for the management of dyslipidaemias: the Task Force for the management of dyslipidaemias of the European Society of Cardiology (ESC) and the European Atherosclerosis Society (EAS). Eur Heart J. 2011 Jul;32(14):1769-818. doi: 10.1093/eurheartj/ehr158. Epub 2011 Jun 28. PMID 21712404
- [Background] Roth EM, McKenney JM, Hanotin C, Asset G, Stein EA. Atorvastatin with or without an antibody to PCSK9 in primary hypercholesterolemia. N Engl J Med. 2012 Nov 15;367(20):1891-900. doi: 10.1056/NEJMoa1201832. Epub 2012 Oct 31. PMID 23113833
- [Background] Soutschek J, Akinc A, Bramlage B, Charisse K, Constien R, Donoghue M, Elbashir S, Geick A, Hadwiger P, Harborth J, John M, Kesavan V, Lavine G, Pandey RK, Racie T, Rajeev KG, Rohl I, Toudjarska I, Wang G, Wuschko S, Bumcrot D, Koteliansky V, Limmer S, Manoharan M, Vornlocher HP. Therapeutic silencing of an endogenous gene by systemic administration of modified siRNAs. Nature. 2004 Nov 11;432(7014):173-8. doi: 10.1038/nature03121. PMID 15538359
- [Background] Stein EA, Mellis S, Yancopoulos GD, Stahl N, Logan D, Smith WB, Lisbon E, Gutierrez M, Webb C, Wu R, Du Y, Kranz T, Gasparino E, Swergold GD. Effect of a monoclonal antibody to PCSK9 on LDL cholesterol. N Engl J Med. 2012 Mar 22;366(12):1108-18. doi: 10.1056/NEJMoa1105803. PMID 22435370
- [Background] Stone NJ, Robinson JG, Lichtenstein AH, Bairey Merz CN, Blum CB, Eckel RH, Goldberg AC, Gordon D, Levy D, Lloyd-Jones DM, McBride P, Schwartz JS, Shero ST, Smith SC Jr, Watson K, Wilson PW, Eddleman KM, Jarrett NM, LaBresh K, Nevo L, Wnek J, Anderson JL, Halperin JL, Albert NM, Bozkurt B, Brindis RG, Curtis LH, DeMets D, Hochman JS, Kovacs RJ, Ohman EM, Pressler SJ, Sellke FW, Shen WK, Smith SC Jr, Tomaselli GF; American College of Cardiology/American Heart Association Task Force on Practice Guidelines. 2013 ACC/AHA guideline on the treatment of blood cholesterol to reduce atherosclerotic cardiovascular risk in adults: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines. Circulation. 2014 Jun 24;129(25 Suppl 2):S1-45. doi: 10.1161/01.cir.0000437738.63853.7a. Epub 2013 Nov 12. No abstract available. PMID 24222016
- [Background] Sullivan D, Olsson AG, Scott R, Kim JB, Xue A, Gebski V, Wasserman SM, Stein EA. Effect of a monoclonal antibody to PCSK9 on low-density lipoprotein cholesterol levels in statin-intolerant patients: the GAUSS randomized trial. JAMA. 2012 Dec 19;308(23):2497-506. doi: 10.1001/jama.2012.25790. PMID 23128163
- [Background] Tabernero J, Shapiro GI, LoRusso PM, Cervantes A, Schwartz GK, Weiss GJ, Paz-Ares L, Cho DC, Infante JR, Alsina M, Gounder MM, Falzone R, Harrop J, White AC, Toudjarska I, Bumcrot D, Meyers RE, Hinkle G, Svrzikapa N, Hutabarat RM, Clausen VA, Cehelsky J, Nochur SV, Gamba-Vitalo C, Vaishnaw AK, Sah DW, Gollob JA, Burris HA 3rd. First-in-humans trial of an RNA interference therapeutic targeting VEGF and KSP in cancer patients with liver involvement. Cancer Discov. 2013 Apr;3(4):406-17. doi: 10.1158/2159-8290.CD-12-0429. Epub 2013 Jan 28. PMID 23358650
- [Background] World Health Organization Cardiovascular Statistics, 2011, http://www.who.int/mediacentre/factsheets/fs317/en/index.html
- [Background] Yusuf S, Hawken S, Ounpuu S, Dans T, Avezum A, Lanas F, McQueen M, Budaj A, Pais P, Varigos J, Lisheng L; INTERHEART Study Investigators. Effect of potentially modifiable risk factors associated with myocardial infarction in 52 countries (the INTERHEART study): case-control study. Lancet. 2004 Sep 11-17;364(9438):937-52. doi: 10.1016/S0140-6736(04)17018-9. PMID 15364185
- [Background] Zhao Z, Tuakli-Wosornu Y, Lagace TA, Kinch L, Grishin NV, Horton JD, Cohen JC, Hobbs HH. Molecular characterization of loss-of-function mutations in PCSK9 and identification of a compound heterozygote. Am J Hum Genet. 2006 Sep;79(3):514-23. doi: 10.1086/507488. Epub 2006 Jul 18. PMID 16909389
- [Background] Zimmermann TS, Lee AC, Akinc A, Bramlage B, Bumcrot D, Fedoruk MN, Harborth J, Heyes JA, Jeffs LB, John M, Judge AD, Lam K, McClintock K, Nechev LV, Palmer LR, Racie T, Rohl I, Seiffert S, Shanmugam S, Sood V, Soutschek J, Toudjarska I, Wheat AJ, Yaworski E, Zedalis W, Koteliansky V, Manoharan M, Vornlocher HP, MacLachlan I. RNAi-mediated gene silencing in non-human primates. Nature. 2006 May 4;441(7089):111-4. doi: 10.1038/nature04688. Epub 2006 Mar 26. PMID 16565705
- [Derived] Dutta S, Shah R, Singhal S, Singh S, Piparva K, Katoch CDS. A systematic review and meta-analysis of tolerability, cardiac safety and efficacy of inclisiran for the therapy of hyperlipidemic patients. Expert Opin Drug Saf. 2024 Feb;23(2):187-198. doi: 10.1080/14740338.2023.2293201. Epub 2023 Dec 19. PMID 38063346
- [Derived] Wright RS, Collins MG, Stoekenbroek RM, Robson R, Wijngaard PLJ, Landmesser U, Leiter LA, Kastelein JJP, Ray KK, Kallend D. Effects of Renal Impairment on the Pharmacokinetics, Efficacy, and Safety of Inclisiran: An Analysis of the ORION-7 and ORION-1 Studies. Mayo Clin Proc. 2020 Jan;95(1):77-89. doi: 10.1016/j.mayocp.2019.08.021. Epub 2019 Oct 17. PMID 31630870
- [Derived] Ray KK, Stoekenbroek RM, Kallend D, Nishikido T, Leiter LA, Landmesser U, Wright RS, Wijngaard PLJ, Kastelein JJP. Effect of 1 or 2 Doses of Inclisiran on Low-Density Lipoprotein Cholesterol Levels: One-Year Follow-up of the ORION-1 Randomized Clinical Trial. JAMA Cardiol. 2019 Nov 1;4(11):1067-1075. doi: 10.1001/jamacardio.2019.3502. PMID 31553410
- [Derived] Leiter LA, Teoh H, Kallend D, Wright RS, Landmesser U, Wijngaard PLJ, Kastelein JJP, Ray KK. Inclisiran Lowers LDL-C and PCSK9 Irrespective of Diabetes Status: The ORION-1 Randomized Clinical Trial. Diabetes Care. 2019 Jan;42(1):173-176. doi: 10.2337/dc18-1491. Epub 2018 Nov 28. PMID 30487231
- [Derived] Ray KK, Stoekenbroek RM, Kallend D, Leiter LA, Landmesser U, Wright RS, Wijngaard P, Kastelein JJP. Effect of an siRNA Therapeutic Targeting PCSK9 on Atherogenic Lipoproteins: Prespecified Secondary End Points in ORION 1. Circulation. 2018 Sep 25;138(13):1304-1316. doi: 10.1161/CIRCULATIONAHA.118.034710. PMID 29735484
- [Derived] Ray KK, Landmesser U, Leiter LA, Kallend D, Dufour R, Karakas M, Hall T, Troquay RP, Turner T, Visseren FL, Wijngaard P, Wright RS, Kastelein JJ. Inclisiran in Patients at High Cardiovascular Risk with Elevated LDL Cholesterol. N Engl J Med. 2017 Apr 13;376(15):1430-1440. doi: 10.1056/NEJMoa1615758. Epub 2017 Mar 17. PMID 28306389

RESULTS

PARTICIPANT FLOW:
Groups:
- Inclisiran 200 mg (Single-dose): 200 mg subcutaneous administration once at Day 1
- Inclisiran 300 mg (Single-dose): 300 mg subcutaneous administration once at Day 1
- Inclisiran 500 mg (Single-dose): 500 mg subcutaneous administration once at Day 1
- Placebo (Single-dose): Saline subcutaneous administration once at Day 1
- Inclisiran 100 mg (Double-dose): 100 mg subcutaneous administration at Day 1 and Day 90
- Inclisiran 200 mg (Double-dose): 200 mg subcutaneous administration at Day 1 and Day 90
- Inclisiran 300 mg (Double-dose): 300 mg subcutaneous administration at Day 1 and Day 90
- Placebo (Double-dose): Saline subcutaneous administration at Day 1 and Day 90
Period: Overall Study
Arm/Group | Inclisiran 200 mg (Single-dose) | Inclisiran 300 mg (Single-dose) | Inclisiran 500 mg (Single-dose) | Placebo (Single-dose) | Inclisiran 100 mg (Double-dose) | Inclisiran 200 mg (Double-dose) | Inclisiran 300 mg (Double-dose) | Placebo (Double-dose)
Started | 60 | 62 | 66 | 65 | 62 | 63 | 61 | 62
Treated | 60 | 61 | 65 | 65 | 61 | 62 | 61 | 62
Completed (LDL-C returned to >80% of baseline from Day 210-360 or completed Day 360 with LDL-C<=80% of baseline) | 59 | 59 | 58 | 60 | 57 | 59 | 57 | 60
Not Completed | 1 | 3 | 8 | 5 | 5 | 4 | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (Single-dose) | Inclisiran 200 mg (Single-dose) | Inclisiran 300 mg (Single-dose) | Inclisiran 500 mg (Single-dose) | Placebo (Double-dose) | Inclisiran 100 mg (Double-dose) | Inclisiran 200 mg (Double-dose) | Inclisiran 300 mg (Double-dose) | Total
Number analyzed (Participants) | 65 | 60 | 62 | 66 | 62 | 62 | 63 | 61 | 501
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 40 | 30 | 27 | 32 | 32 | 24 | 37 | 31 | 253
  >=65 years | 25 | 30 | 35 | 34 | 30 | 38 | 26 | 30 | 248
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (11.4) | 63.9 (10.8) | 64.1 (12.8) | 62.1 (12.4) | 62.8 (10.3) | 65.2 (9.4) | 62.3 (10.8) | 64.1 (9.4) | 63.6 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 20 | 19 | 29 | 23 | 24 | 16 | 175
  Male | 42 | 39 | 42 | 47 | 33 | 39 | 39 | 45 | 326
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 3 | 1 | 2 | 2 | 6 | 4 | 29
  Not Hispanic or Latino | 58 | 56 | 59 | 65 | 60 | 60 | 57 | 57 | 472
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 1 | 0 | 2 | 0 | 1 | 6
  Asian | 0 | 2 | 2 | 2 | 1 | 1 | 0 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 4 | 4 | 2 | 0 | 3 | 2 | 2 | 1 | 18
  White | 59 | 53 | 56 | 63 | 58 | 57 | 61 | 58 | 465
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 8 | 8 | 7 | 12 | 10 | 10 | 7 | 9 | 71
  Netherlands | 22 | 21 | 21 | 21 | 20 | 20 | 23 | 21 | 169
  United States | 12 | 10 | 10 | 12 | 8 | 10 | 12 | 10 | 84
  United Kingdom | 11 | 11 | 11 | 11 | 10 | 9 | 11 | 12 | 86
  Germany | 12 | 10 | 13 | 10 | 14 | 13 | 10 | 9 | 91

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in LDL-C From Baseline to Day 180
Description: Percent Change in LDL-C (beta-quantification) from Baseline to Day 180 in MITT Population
Time Frame: Baseline to 180 days
Population: Modified intent-to-treat (MITT) population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Groups:
- Placebo (Single Dose): Saline via subcutaneous injection - Single Dose on Day 1
- 200 mg (Single Dose): 200 mg Inclisiran via subcutaneous injection - Single Dose on Day 1
- 300 mg (Single Dose): 300 mg Inclisiran via subcutaneous injection - Single Dose on Day 1
- 500 mg (Single Dose): 500 mg Inclisiran via subcutaneous injection - Single Dose on Day 1
- Placebo (Double Dose): Saline via subcutaneous injection - Two Doses: Day 1 and Day 90
- 100 mg (Double Dose): 100 mg Inclisiran via subcutaneous injection - Two Doses: Day 1 and Day 90
- 200 mg (Double Dose): 200 mg Inclisiran via subcutaneous injection - Two Doses: Day 1 and Day 90
- 300 mg (Double Dose): 300 mg Inclisiran via subcutaneous injection - Two Doses: Day 1 and Day 90
Arm/Group | Placebo (Single Dose) | 200 mg (Single Dose) | 300 mg (Single Dose) | 500 mg (Single Dose) | Placebo (Double Dose) | 100 mg (Double Dose) | 200 mg (Double Dose) | 300 mg (Double Dose)
Number analyzed (Participants) | 64 | 60 | 60 | 60 | 61 | 59 | 60 | 59
Percent change | 2.1 [-2.9 to 7.2] | -27.9 [-33.1 to -22.7] | -38.4 [-43.6 to -33.2] | -41.9 [-47.2 to -36.7] | 1.8 [-2.6 to 6.3] | -35.5 [-40.0 to -31.0] | -44.9 [-49.3 to -40.4] | -52.6 [-57.1 to -48.1]
Statistical Analysis 1: Comparison: Placebo (Single Dose) vs 200 mg (Single Dose); Test type: Superiority — Two sample t-tests were performed to test the superiority of any dosing group over placebo. A Dunnett multiple t-test procedure was applied to adjust for multiple comparisons with six different dosing regimens; p < 0.0001, t-test, 1 sided — This P-Value applies to the comparison of the mean percent change at Day 180 for the 200 mg (Single-Dose) Inclisiran group versus Placebo (Single-Dose)
Statistical Analysis 2: Comparison: Placebo (Single Dose) vs 300 mg (Single Dose); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, t-test, 1 sided — This P-Value applies to the comparison of the mean percent change at Day 180 for the 300 mg (Single-Dose) Inclisiran group versus Placebo (Single-Dose)
Statistical Analysis 3: Comparison: Placebo (Single Dose) vs 500 mg (Single Dose); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, t-test, 1 sided — This P-Value applies to the comparison of the mean percent change at Day 180 for the 500 mg (Single-Dose) Inclisiran group versus Placebo (Single-Dose)
Statistical Analysis 4: Comparison: Placebo (Double Dose) vs 100 mg (Double Dose); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, t-test, 1 sided — This P-Value applies to the comparison of the mean percent change at Day 180 for the 100 mg Double-Dose) Inclisiran group versus Placebo (Double-Dose)
Statistical Analysis 5: Comparison: Placebo (Double Dose) vs 200 mg (Double Dose); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, t-test, 1 sided — This P-Value applies to the comparison of the mean percent change at Day 180 for the 200 mg Double-Dose) Inclisiran group versus Placebo (Double-Dose)
Statistical Analysis 6: Comparison: Placebo (Double Dose) vs 300 mg (Double Dose); Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, t-test, 1 sided — This P-Value applies to the comparison of the mean percent change at Day 180 for the 300 mg Double-Dose) Inclisiran group versus Placebo (Double-Dose)

2. Secondary Outcome: Percentage Change in LDL-C From Baseline to Day 90
Description: Percent Change in LDL-C (beta-quantification) from Baseline to Day 90 in MITT Population
Time Frame: Baseline to 90 days
Population: In this analysis, the single and double-dose 200mg arms were combined, as were the single and double-dose 300mg arms. The second dose for patients in double-dose arms was given on Day 90. Therefore, up to day 90, those patients in double-dose arms received the same treatment as patients in the single dose arms within the same dose amount.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent change
Groups:
- Single Dose 500 mg: 500 mg subcutaneous injection - Single Dose on Day 1 (2 injections)
- Double Dose 100 mg: 200 mg Inclisiran via subcutaneous injection - Two Doses (Day 1 and Day 90)
- Single and Double Dose Placebo: Saline: Single Dose (Day 1) or Two Doses (Day 1 and Day 90)
- Single and Double Dose 200 mg: 200 mg Inclisiran via subcutaneous injection: Single Dose (Day 1) or Two Doses (Day 1 and Day 90)
- Single and Double Dose 300 mg: 300 mg Inclisiran via subcutaneous injection: Single Dose (Day 1) or Two Doses (Day 1 and Day 90)
Arm/Group | Single Dose 500 mg | Double Dose 100 mg | Single and Double Dose Placebo | Single and Double Dose 200 mg | Single and Double Dose 300 mg
Number analyzed (Participants) | 60 | 59 | 125 | 120 | 118
Percent change | -49 [-53.8 to -44.2] | -34.2 [-39.1 to -29.3] | -0.8 [-4.2 to 2.5] | -41.8 [-45.3 to -38.4] | -45.7 [-49.2 to -42.3]

3. Secondary Outcome: Percent Change From Baseline In LDL-C Levels At Day 60, Day 120, and Day 210
Description: This outcome measure evaluated the effects of both single- and double-dose inclisiran on LDL-C levels in the mITT population from baseline to Day 60, Day 120, and Day 210.
Time Frame: Baseline, Day 60, Day 120, and Day 210
Measure: Mean (95% Confidence Interval); unit: Percent change
Groups:
- Placebo (Single Dose): Saline subcutaneous administration once at Day 1
- Inclisiran 200 mg (Single Dose): 200 mg subcutaneous administration once at Day 1
- Inclisiran 300 mg (Single Dose): 300 mg subcutaneous administration once at Day 1
- Inclisiran 500 mg (Single Dose): 500 mg subcutaneous administration once at Day 1
- Placebo (Double Dose): Saline subcutaneous administration twice at Day 1 and Day 90
- Inclisiran 100 mg (Double Dose): 100 mg subcutaneous administration twice at Day 1 and Day 90
- Inclisiran 200 mg (Double Dose): 200 mg subcutaneous administration twice at Day 1 and Day 90
- Inclisiran 300 mg (Double Dose): 300 mg subcutaneous administration twice at Day 1 and Day 90
Arm/Group | Placebo (Single Dose) | Inclisiran 200 mg (Single Dose) | Inclisiran 300 mg (Single Dose) | Inclisiran 500 mg (Single Dose) | Placebo (Double Dose) | Inclisiran 100 mg (Double Dose) | Inclisiran 200 mg (Double Dose) | Inclisiran 300 mg (Double Dose)
Number analyzed (Participants) | 64 | 60 | 60 | 60 | 61 | 59 | 60 | 59
Percent change
  Day 60 | -4.27 [-7.84 to -0.7] | -44.32 [-50.55 to -38.09] | -50.87 [-55.62 to -46.12] | -49.58 [-54.12 to -45.04] | -1.92 [-6.7 to 2.85] | -35.73 [-40.23 to -31.23] | -44.28 [-49.1 to -39.47] | -50.99 [-55.51 to -45.67]
  Day 120 | -0.91 [-5.17 to 3.34] | -36.94 [-42.8 to -31.08] | -43.32 [-48.95 to -37.68] | -46.42 [-50.63 to -42.22] | 0.17 [-3.61 to 3.95] | -41.37 [-45.94 to -36.8] | -49.54 [-54.6 to -44.49] | -54.73 [-59.88 to -49.58]
  Day 210 | 1.45 [-3.61 to 6.06] | -28.98 [-36.83 to -21.12] | -35.39 [-41.47 to -29.31] | -39.2 [-43.71 to -34.68] | 0.58 [-4.58 to 5.74] | -31.67 [-36.08 to -27.27] | -42.59 [-47.11 to -38.08] | -50.54 [-54.83 to -46.25]

4. Secondary Outcome: Number of Participants With an LDL-C Greater Than 80% of the Baseline Value at Day 180 and Day 210
Description: This outcome measure evaluated the number of participants (single and double dose) in the mITT population with an LDL-C greater than 80% of the baseline value at Day 180 and Day 210.
Time Frame: Baseline, Day 180, Day 210
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Single-dose) | Inclisiran 200 mg (Single-dose) | Inclisiran 300 mg (Single-dose) | Inclisiran 500 mg (Single-dose) | Placebo (Double-dose) | Inclisiran 100 mg (Double-dose) | Inclisiran 200 mg (Double-dose) | Inclisiran 300 mg (Double-dose)
Number analyzed (Participants) | 64 | 60 | 60 | 60 | 61 | 59 | 60 | 59
Participants
  Day 180 | 35 | 6 | 5 | 0 | 29 | 2 | 1 | 0
  Day 210 | 34 | 8 | 5 | 2 | 34 | 1 | 1 | 1

5. Secondary Outcome: Number of Participants With Individual Responsiveness as Measured By LDL-C Levels at Day 90 and Day 180
Description: This outcome measure evaluated the individual responsiveness of participants to inclisiran (single and double dose) in the mITT population as defined by an LDL-C level of <25 mg/deciliter [dL] at Day 90 and Day 180.
Time Frame: Day 90, Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Single-dose) | Inclisiran 200 mg (Single-dose) | Inclisiran 300 mg (Single-dose) | Inclisiran 500 mg (Single-dose) | Placebo (Double-dose) | Inclisiran 100 mg (Double-dose) | Inclisiran 200 mg (Double-dose) | Inclisiran 300 mg (Double-dose)
Number analyzed (Participants) | 64 | 60 | 60 | 60 | 61 | 59 | 60 | 59
Participants
  Day 90 | 0 | 0 | 5 | 3 | 0 | 0 | 1 | 0
  Day 180 | 0 | 0 | 1 | 2 | 0 | 1 | 2 | 3

6. Secondary Outcome: Number of Participants With Greater Or Equal To 50% LDL-C Reduction From Baseline At Day 180
Description: This outcome measure evaluated the number of participants (single and double dose) in the mITT population with an LDL-C reduction greater than 50% of the baseline value at Day 180.
Time Frame: Baseline, Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Single-dose) | Inclisiran 200 mg (Single-dose) | Inclisiran 300 mg (Single-dose) | Inclisiran 500 mg (Single-dose) | Placebo (Double-dose) | Inclisiran 100 mg (Double-dose) | Inclisiran 200 mg (Double-dose) | Inclisiran 300 mg (Double-dose)
Number analyzed (Participants) | 64 | 60 | 60 | 60 | 61 | 59 | 60 | 59
Participants | 0 | 9 | 19 | 16 | 0 | 14 | 27 | 32

7. Secondary Outcome: Percentage Change in PCSK9 Levels From Baseline at Day 180
Description: This outcome measure evaluated the percent change in proprotein convertase subtilisin/kexin type 9 (PCSK9) from baseline to Day 180 in participants (single and double dose) in the mITT population.
Time Frame: Baseline, Day 180
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (Single Dose) | Inclisiran 200 mg (Single Dose) | Inclisiran 300 mg (Single Dose) | Inclisiran 500 mg (Single Dose) | Placebo (Double Dose) | Inclisiran 100 mg (Double Dose) | Inclisiran 200 mg (Double Dose) | Inclisiran 300 mg (Double Dose)
Number analyzed (Participants) | 64 | 60 | 60 | 60 | 61 | 59 | 60 | 59
percent change | 2.2 (23.4) | -47.9 (21) | -56 (19.2) | -59.3 (18) | -1.2 (20.7) | -53.2 (20.9) | -66.2 (15.6) | -69.1 (12.1)

8. Secondary Outcome: Percentage Change in Other Lipids and Apolipoproteins From Baseline to Day 180
Description: This outcome measure evaluated the percent change from baseline to Day 180 in cholesterol (total, high-density lipoprotein [HDL], non-HDL) and apolipoproteins (B, A1) in participants (single and double dose) in the mITT population.
Time Frame: Baseline, Day 180
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo (Single Dose) | Inclisiran 200 mg (Single Dose) | Inclisiran 300 mg (Single Dose) | Inclisiran 500 mg (Single Dose) | Placebo (Double Dose) | Inclisiran 100 mg (Double Dose) | Inclisiran 200 mg (Double Dose) | Inclisiran 300 mg (Double Dose)
Number analyzed (Participants) | 64 | 60 | 60 | 60 | 61 | 59 | 60 | 59
percent change
  Total Cholesterol | 1.8 (12.1) | -17.6 (19) | -23.7 (15.7) | -26.6 (10.7) | 0.7 (12.3) | -22.4 (12.4) | -26.8 (13) | 33.2 (11.3)
  Non-HDL Cholesterol | 1.5 (16.7) | -25.1 (26.3) | -35.2 (20.2) | -36.9 (14) | 1.3 (16.9) | -31.7 (15.1) | -38.9 (16.8) | -46 (14.6)
  HDL Cholesterol | 3.8 (15.6) | 4.4 (14.8) | 8.8 (11.1) | 6.9 (14) | 0.5 (12.5) | 7.6 (12.2) | 10.3 (15.3) | 8.6 (14.9)
  Apolipoprotein B | 1.7 (14.7) | -22.9 (21) | -30.8 (18) | -33.1 (12.7) | 0.9 (13) | -27.8 (13.4) | -35 (15.8) | -40.9 (14.8)
  Apolipoprotein A1 | 3.6 (10.6) | 2.9 (9.3) | 3.8 (8.9) | 4.1 (10.9) | 0.8 (8.3) | 5.5 (10.6) | 8.6 (11.5) | 6.2 (11.9)

9. Secondary Outcome: Number of Participants Who Attained Global Lipid Modification Targets for Level of Atherosclerotic Cardiovascular Disease Risk
Description: This outcome measure evaluated the proportion of participants (single and double dose) in the mITT population who attained a global lipid modification target by baseline cardiovascular risk group, looking specifically at LDL-C levels (mg/dL) in the category of cardiovascular disease (CVD).
  CVD was defined as a participant who had at least 1 of the following: prior myocardial infarction, prior percutaneous coronary intervention, prior coronary artery bypass graft, prior stroke, prior transient ischemic attack, peripheral artery disease.
Time Frame: Baseline, Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Single-dose) | Inclisiran 200 mg (Single-dose) | Inclisiran 300 mg (Single-dose) | Inclisiran 500 mg (Single-dose) | Placebo (Double-dose) | Inclisiran 100 mg (Double-dose) | Inclisiran 200 mg (Double-dose) | Inclisiran 300 mg (Double-dose)
Number analyzed (Participants) | 64 | 60 | 60 | 60 | 61 | 59 | 60 | 59
Participants
  CVD | 45 | 43 | 46 | 33 | 45 | 41 | 39 | 42
  <70 mg/dL | 0 | 16 | 27 | 18 | 1 | 24 | 27 | 33

10. Secondary Outcome: Percentage Change in Other Lipids and Inflammatory Markers From Baseline to Day 180
Description: This outcome measure evaluated the percent change from baseline to Day 180 in triglycerides, very-low-density lipoprotein (VLDL) cholesterol, lipoprotein(a), and high sensitivity C-reactive protein (hsCRP) in participants (single and double dose) in the mITT population.
Time Frame: Baseline, Day 180
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Placebo (Single Dose) | Inclisiran 200 mg (Single Dose) | Inclisiran 300 mg (Single Dose) | Inclisiran 500 mg (Single Dose) | Placebo (Double Dose) | Inclisiran 100 mg (Double Dose) | Inclisiran 200 mg (Double Dose) | Inclisiran 300 mg (Double Dose)
Number analyzed (Participants) | 64 | 60 | 60 | 60 | 61 | 59 | 60 | 59
percent change
  Triglycerides | 6.4 [-15.9 to 21.9] | 1.1 [-18.5 to 17.8] | -12.8 [-27.8 to 7.8] | -12.2 [-25.6 to 7.7] | -3 [-17.2 to 22.6] | -6.3 [-17.6 to 10.9] | 0.7 [-22.4 to 11.3] | -14.2 [-26.4 to 5.4]
  VLDL Cholesterol | 2.4 [-30.7 to 30.5] | -11.6 [-35.8 to 23.3] | -23.8 [-43 to -6.4] | -14.6 [-34.8 to 3.5] | 2.7 [-20 to 26.7] | -16.4 [-31.3 to 0] | -21.2 [-38.5 to 13.2] | -16 [-38.2 to 9.1]
  Lipoprotein(a) | 0.5 [-13.9 to 14.8] | -14.3 [-29.5 to -3.5] | -14.3 [-25.4 to -5.6] | -18.2 [-35 to 1.6] | 0 [-10 to 12.4] | -14.9 [-26.2 to -1.9] | -17.3 [-31.9 to -7.7] | -25.6 [-38.5 to -15.2]
  hsCRP | -5.3 [-40.8 to 28.4] | 7.1 [-30.7 to 70.9] | -16.2 [-45.8 to 50] | -19.8 [-50 to 32.7] | -20 [-50 to 30] | -12.5 [-42.9 to 29.4] | -16.3 [-34.6 to 24.3] | -16.7 [-50.9 to 33.3]

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events up to Day 360
Arm/Group | Placebo (Single Dose) | Inclisiran 200 mg (Single Dose) | Inclisiran 300 mg (Single Dose) | Inclisiran 500 mg (Single Dose) | Placebo (Double Dose) | Inclisiran 100 mg (Double Dose) | Inclisiran 200 mg (Double Dose) | Inclisiran 300 mg (Double Dose)
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/60 | 0/61 | 1/65 | 0/62 | 0/61 | 1/62 | 0/61
Serious Adverse Events (participants affected / at risk) | 3/65 | 11/60 | 11/61 | 8/65 | 7/62 | 13/61 | 8/62 | 9/61
Other Adverse Events (participants affected / at risk) | 50/65 | 49/60 | 49/61 | 54/65 | 51/62 | 47/61 | 49/62 | 51/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Single Dose) (N=65) | Inclisiran 200 mg (Single Dose) (N=60) | Inclisiran 300 mg (Single Dose) (N=61) | Inclisiran 500 mg (Single Dose) (N=65) | Placebo (Double Dose) (N=62) | Inclisiran 100 mg (Double Dose) (N=61) | Inclisiran 200 mg (Double Dose) (N=62) | Inclisiran 300 mg (Double Dose) (N=61)
Anameia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Atriventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aorta-oesophageal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
large instestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Proctitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Volvulus (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Device dislocation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Srent-graft endoleak (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vascular stent restenosis (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Implant site infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Listeria sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Osteomyelitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Wound abcess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Limb crushing injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Upperlimb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weaning failure (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle necrosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Adeoncarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bladder transitional cell carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Non-small cell lung cancer stage 1 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tongue neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lacunar stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Spinal cord ischaemia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Calculus urinary (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Stress urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aortic dissection (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Intermittent claudication (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Single Dose) (N=65) | Inclisiran 200 mg (Single Dose) (N=60) | Inclisiran 300 mg (Single Dose) (N=61) | Inclisiran 500 mg (Single Dose) (N=65) | Placebo (Double Dose) (N=62) | Inclisiran 100 mg (Double Dose) (N=61) | Inclisiran 200 mg (Double Dose) (N=62) | Inclisiran 300 mg (Double Dose) (N=61)
Angina pectoris (Cardiac disorders) | 1 | 2 | 4 | 1 | 2 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 3 | 2 | 0 | 3 | 2 | 1 | 4
Constipation (Gastrointestinal disorders) | 1 | 4 | 2 | 1 | 2 | 0 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 4 | 4 | 2 | 3 | 7 | 5
Nausea (Gastrointestinal disorders) | 2 | 1 | 1 | 4 | 3 | 2 | 4 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 4 | 0
Fatigue (General disorders) | 5 | 2 | 4 | 2 | 6 | 2 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 3 | 2 | 1 | 2 | 3 | 1 | 1
Influenza (Infections and infestations) | 3 | 3 | 4 | 5 | 2 | 3 | 4 | 5
Nasopharyngitis (Infections and infestations) | 4 | 8 | 9 | 9 | 8 | 8 | 5 | 11
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 4 | 5 | 2 | 2 | 1 | 3
Urinary tract infection (Infections and infestations) | 1 | 1 | 5 | 0 | 4 | 1 | 1 | 2
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 2 | 5 | 3 | 1 | 2
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1 | 1 | 4 | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 3 | 1 | 1 | 0 | 5 | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 4 | 4 | 4 | 1 | 2 | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 4 | 4 | 4 | 2 | 6 | 1 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 1 | 4 | 0 | 0 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 6 | 3 | 3 | 7 | 5 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 2 | 1 | 2 | 4 | 1 | 4 | 1
Dizziness (Nervous system disorders) | 3 | 1 | 2 | 2 | 6 | 3 | 3 | 3
Headache (Nervous system disorders) | 6 | 2 | 2 | 2 | 5 | 5 | 1 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 7 | 3 | 3 | 1 | 6 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 0 | 1 | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 2 | 3 | 1 | 3 | 4 | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that Sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period of more than 60 days but less than/equal to 180 days from the time submitted to Sponsor for review, allowing Sponsor to file a patent application or take such other measures as Sponsor deems appropriate to establish and preserve its proprietary rights. Sponsor may remove confidential or proprietary information.

DOCUMENTS (2):
  • Study Protocol (2016-04-12): https://cdn.clinicaltrials.gov/large-docs/27/NCT02597127/Prot_000.pdf
  • Statistical Analysis Plan (2016-01-11): https://cdn.clinicaltrials.gov/large-docs/27/NCT02597127/SAP_001.pdf